CLINICAL TRIAL: NCT01476098
Title: Two Part Study to Investigate Pharmacokinetics (PK) & Pharamcodynamics (PD) of SB-705498 in Cough. Part A:Open Label Study in Healthy Subjects to Determine Exposure to SB-705498. Part B:Double-blind, Placebo Controlled, Cross Over Study to Investigate Effect of SB-705498 on Capsaicin Induced Cough and 24 Hour Cough Counts in Cough Patients
Brief Title: A Study to Investigate the Effect of SB-705498 on Chronic Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 114693
Record Dates: First submitted 2011-10-13; First posted 2011-11-22 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — SB 705498

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Placebo Comparator): incremental doses capsaicin
  Interventions: Drug: Placebo; Drug: SB-705498
- Arm 2 (Active Comparator): incremenrtal doses casaicin
  Interventions: Drug: Placebo; Drug: SB-705498

INTERVENTIONS:
Drug: Placebo — SB-705498 placebo
Drug: SB-705498 — 400 or 600mg oral SB-705498

SUMMARY:
This study is designed to loook at the affect of oral SB-705498 on cough following an inhaled capsaicin challenge

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 30 -75 (Part A) and 18-75 (Part B) years of age inclusive.
* Non-child bearing women or women of child bearing potential if they agree to use contraception as indicated by the protocol
* Non-smoker for at least 6 months with a pack history <5 pack years (Pack years = (No. of cigarettes smoked/day/20) x No. of years smoked).
* Body weight > 50 kg and body mass index (BMI) within the range 19 - 30.0 kg/m2 (inclusive).
* Capable of giving written informed consent.
* Agree to use contraception listed as acceptable
* Normal 12-lead ECG at screening.
* Chronic cough (Part B only)
* Good general health, apart from chronic cough (part B only), as determined by a responsible physician.

Exclusion Criteria:

* A history of gastrointestinal, hepatic, renal or multiple cardiovascular risk factors.
* Positive pre-study drug/alcohol screen.
* Positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for human immunodeficiency virus (HIV) antibody (if determined by the local standard operating procedures (SOPs)).
* History of regular alcohol consumption within 6 months of the study.
* Exposure to more than four new chemical entities within 12 months prior to the start of the study.
* Participation in a clinical trial with a new molecule entity or any other clinical trial within 30 days of the start of the study.
* Use of prescription or non-prescription drugs, as well as of vitamins, herbal and dietary supplements (including St John's Wort) within 7 days prior to study.
* known history of lung cancer
* current treatment with oral corticosteriods or other immunosupressive agents
* FEV1 less than 80% of predicted value at screening
* Any subject who does not reach C5 following 250uM oral capsaicin
* History of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation.
* Donation of blood or blood products in excess of 500mL within a 56 day period prior the start study.
* Pregnant females as determined by positive serum or urine human chorionic gonadotropin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of area under the plasma concentration-time curve from time zero to 4 hours AUC(0-4) and from time zero (pre-dose) to last time of quantifiable concentration AUC(0-t)- Part A | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 10 hours post-dose
  AUC(0-4) is a measure of the average amount of study drug in the blood plasma over a period of 4 hours after the dose and AUC(0-t) is a measure average amount of study drug in the blood plasma over a period of last time of quantifiable concentration. Both the parameters were calculated by standard non-compartmental analysis. Blood samples for PK analysis were obtained at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 10 hours post-dose.
Maximum observed concentration (Cmax) following 10 hour sampling of a single dose of SB-705498 - Part A | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 10 hours post-dose Day 1
  Cmax is defined as the maximum or "peak" concentration of a drug observed after its administration. Cmax is one of the parameters of particular use in estimating the bioavailability of drugs, by measuring the total amount of drug absorbed. It was calculated by standard non-compartmental analysis. Blood samples for PK analysis were obtained at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 10 hours post-dose.
Time of occurrence of Cmax (Tmax) following 10 hour sampling of a single dose of SB-705498 -Part A | pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 10 hours post-dose
  Tmax is defined as the time of occurrence of Cmax. Blood samples for PK analysis were obtained at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 10 hours post-dose.
Capsaicin concentration required to achieve Five or more coughs (C5) following a single dose of SB-705498 at Tmax as compared to baseline- Part A | Day -1 (baseline) and Day 1 (2 hours post dose
  The concentration of capsaicin required to elicit 5 coughs was analyzed. The distributional properties were investigated, and the endpoint was logged (base 2) for analysis and the difference from Day -1 (baseline) was taken (equivalent to ratio on log scale).
Capsaicin concentration required to achieve C5 following a single dose of SB-705498 or placebo- Part B | Day -1, Day 1 (2hrs and 24 hrs post dose)
  The concentration of capsaicin required to elicit 5 coughs was analyzed. The distributional properties were investigated, and the endpoint was logged (base 2) for analysis and the difference from Day -1 (baseline) was taken (equivalent to ratio on log scale).
Cough Count Per 24 hour following single dose of SB-705498 as compared to placebo- Part B | Day -1 and Day 1 (2 and 24 hours)
  24 hour cough count (rate/h) following single dose of SB-705498 as compared to placebo were analyzed by first log transforming the cough counts taken on Day -1 and on Day 1 of each period in the 24 hours post dose. The cough count rates were log(10) transformed.

SECONDARY OUTCOMES:
Capsaicin concentration required to achieve two or more coughs (C2) following a single dose of SB-705498 at Tmax as compared to baseline- Part A | Day -1 and Day 1 (2 hours post dose)
  The concentration of capsaicin required to elicit 2 coughs was analyzed. The distributional properties were investigated, and the endpoint was logged (base 2) for analysis and the difference from Day -1 (baseline) was taken (equivalent to ratio on log scale).
Capsaicin concentration required to achieve C2 following a single dose of SB-705498 at Tmax as compared to baseline- Part B | Day 1 (2 and 24 hours post dose)
Changes in the Cough Quality of Life Questionnaire (CQLQ) following a single dose of SB-705498 compared to placebo- Part B | Day -1 and 14
  It is a validated, 28-item assessment tool designed to evaluate decrements in quality of life due to chronic cough. This questionnaire measures cough-related symptoms, as well as the social implications and psychological impact. Examples of items include, "I cannot sleep at night" and "I cough and it makes me retch." The final score is obtained by summing the responses to 28 questions, each scored on a 1-4 scale, where 1 is "strongly disagree," and 4 is "strongly agree." The minimum and maximum CQLQ scores are 28 and 112 respectively, with increasing score indicating more severe impairment.
Urge to cough Visual Analogue Scale (VAS) following single dose of SB-705498- Part B | Day -1 and Day 1 (pre-dose 2 and 24 hours)
  VAS following single dose of SB-705498 was summarized on Day -1, and Day 1 pre-dose, 2 and 24 hours.
Capsaicin concentration required to achieve C5 following a single dose of SB-705498 at 24 hours as compared to baseline-Part B | Day -1 and Day 1 (2 and 24 hours post dose)
  The concentration of capsaicin required to elicit 5 coughs was analyzed. The distributional properties were investigated, and the endpoint was logged (base 2) for analysis and the difference from Day -1 (baseline) was taken (equivalent to ratio on log scale).
Capsaicin concentration required to achieve C2 following a single dose of SB-705498 at 24 hours as compared to baseline- Part B | Day -1 and Day 1 (2 and 24 hours post dose)
  The concentration of capsaicin required to elicit 2 coughs was analyzed. The distributional properties were investigated, and the endpoint was logged (base 2) for analysis and the difference from Day -1 (baseline) was taken (equivalent to ratio on log scale).
The 24-hour cough count (rate) subdivided by day and night cough counts (rates) to give day/night specific values by treatment group-Part B | Up to Day 2 (Period 2)
  Different cough intervals were investigated, such as a day and night time rate. Participants were treated as a random effect in the model. The mean treatment difference and associated 95% confidence interval was back-transformed to provide a treatment ratio and 95% confidence interval for the ratio.
Number participants with Adverse Events(AEs) and serious adverse events (SAEs)- Part A | Up to Day 7
  An adverse event (AE) was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Number participants with AEs and SAEs- Part B | up to Day 42
  An adverse event (AE) was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started. An adverse event was therefore any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Summary of vital signs -systolic and diastolic blood pressure (Part A) | Up to Day 7
  Systolic and diastolic blood pressure was assessed on pre dose and 2, 10 hours post dose.
Summary of vital signs -systolic and diastolic blood pressure (Part B) | Up to Day 42
  Systolic and diastolic blood pressure was assessed on pre dose and 4 hours post dose.
Summary of Vital Signs- Heart rate (Part A) | Up to Day 7
  Heart rate was assessed on pre dose and 2, 10 hours post dose.
Summary of Vital Signs- Heart rate (Part B) | Up to Day 42
  Heart rate was assessed on pre dose and 4 hours post dose.
Summary of Vital Signs- Body temperature (Part A) | Up to Day 7
  Body temperature was measured with a tympanic thermometer at pre-dose, 1, 2, 4, 10 hours post dose.
Summary of Vital Signs- Body temperature (Part B) | Up to Day 42
  Body temperature was measured with a tympanic thermometer at pre-dose, 1, 2, 4, 24 hours post dose.
Number of participants with ECG findings- Part A | Up to Day 7
  Single 12-lead ECGs was obtained at each time point during the study using an ECG machine. Participants with abnormal values have been presented.
Number of participants with ECG findings- Part B | Up to Day 42
  Single 12-lead ECGs was obtained at each time point during the study using an ECG machine. Participants with abnormal values have been presented.
Number of participants with potential clinical importance (PCI) laboratory assessments- hematology Part A | Up to 4 weeks
  Hematology PCI values were: White Blood Cell Count; 0.67 (low) and 1.82 (high), Neutrophil Count; 0.83 (low), Hemoglobin (male); 1.03 (high), Hemoglobin (female); 1.13 (high), Hematocrit (male); 1.02 (high), Hematocrit (female); 1.17(high), Platelet Count; 0.67 and 1.57 (high), Lymphocytes; 0.81 (low).
Number of participants with potential clinical importance (PCI) laboratory assessments- hematology Part B | Up to 13 weeks
  Hematology PCI values were: White Blood Cell Count; 0.67 (low) and 1.82 (high), Neutrophil Count; 0.83 (low), Hemoglobin (male); 1.03 (high), Hemoglobin (female); 1.13 (high), Hematocrit (male); 1.02 (high), Hematocrit (female); 1.17(high), Platelet Count; 0.67 and 1.57 (high), Lymphocytes; 0.81 (low).
Number of participants with potential clinical importance (PCI) laboratory assessments- clinical biochemistry Part A | Up to 4 weeks
  Clinical biochemistry PCI values were: Albumin; 0.86 (low), Calcium; 0.91(low) and 1.06 (high), Glucose; 0.71 (low) and 1.41 (high), Potassium; 0.86 (low) and 1.10 (high), Sodium; 0.96(low) and 1.03(high).
Number of participants with potential clinical importance (PCI) laboratory assessments- clinical biochemistry Part B | Up to 13 weeks
  Clinical biochemistry PCI values were: Albumin; 0.86 (low), Calcium; 0.91(low) and 1.06 (high), Glucose; 0.71 (low) and 1.41 (high), Potassium; 0.86 (low) and 1.10 (high), Sodium; 0.96(low) and 1.03(high).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114693 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register